CLINICAL TRIAL: NCT04744064
Title: Influence of Protein and Carbohydrate Ingestion on Health Related Adaptations to Recreational Soccer - a Randomized Controlled Trial
Brief Title: Soccer Training and Influence of Protein and Carbohydrate Ingestion on Health
Acronym: SPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Jonas Tybirk, Research Assistent, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Soccer and health
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Healthy
MeSH Terms: interventions — Proteins; Carbohydrates

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Soccer and protein supplementation (Experimental): Soccer training and post exercise supplementation of protein enriched beverage
  Interventions: Dietary Supplement: Protein and carbohydrate
- Soccer and carbohydrate supplementation (Experimental): Soccer training and post exercise supplementation of carbohydrate enriched beverage
  Interventions: Dietary Supplement: Protein and carbohydrate
- Control group (No Intervention): A preliminary control group continueing normal lifestyle

INTERVENTIONS:
Dietary Supplement: Protein and carbohydrate — Intake of 2 x 250 ml of either protein (750 KJ, 21.0 g protein (milk protein), 15.0 g carbohydrate, 4.5 g fat ) or carbohydrate ( 750 KJ, 0 g protein, 0 g fat and 49.2 g carbohydrate (2:1 ratio of maltodextrin: fructose))
  Other Names: Arla Foods Amba, Viby Denmark and Maxim Sports Drink, Orkla Health A/S, Ishøj Denmark
  Arms: Soccer and carbohydrate supplementation; Soccer and protein supplementation

SUMMARY:
The aim of the study was to examine the adaptive response to recreational soccer, conducted as small-sided games, and the effect of supplementing with either protein or carbohydrate after each training session in 10 weeks.

One hundred fifty one middle-aged women and men were randomized into a group ingesting protein or carbohydrate beverages immediately after recreational soccer and prior to bedtime on training days or a control group maintained their normal activities. Training was performed 2.1 times per week for 10 weeks.

DETAILED DESCRIPTION:
We hypothesized that recreational soccer training followed by protein supplementation would have superior beneficial effects on body composition and health compared to recreational soccer training followed by carbohydrate supplementation. The aim of the present study was to examine the effects of ingesting beverages rich in either protein or carbohydrate during a 10-week recreational soccer training period on the adaptive response of lean body mass (primary outcome parameter), fat mass, bone mass density, fitness and health related blood markers in untrained women and men.

Three-hundred-twenty-nine middle-aged men and women were enrolled. One-hundred-fifty-one meet the inclusion criteria and were randomized to two soccer training groups with supplementation of either protein enriched (PG) or carbohydrate enriched (CG) beverages. Prior to the intervention period forty-four of these subjects (18 women and 26 men) completed testing before and after a 10-week period (CON).

The study was a double-blinded experiment. All subjects in the training groups were offered three training sessions per week. Average attendance were 2.1 sessions per week in both PG and CG. Each session lasted around 1 h and was initiated with low to moderate intensity warming for 10 min followed by small-sided (4v4 up to 7v7) soccer matches with a duration of five min separated by 1-2 min of recovery. The subjects in PG and CG ingested a drink of 250 ml immediately after completion of training sessions and again in the evening before bedtime. Subjects in PG ingested per serving a protein enriched milk-based beverage containing in total 750 KJ, 21.0 g protein (milk protein), 15.0 g carbohydrate, 4.5 g fat. Subjects in CG ingested per serving an isocaloric carbohydrate-rich beverage containing in total 750 KJ, 0 g protein, 0 g fat and 49.2 g carbohydrate (2:1 ratio of maltodextrin: fructose). Before the intervention, the participants completed a weighed dietary record on three consecutive days, including one weekend day. During week five or six in INT, a weighed dietary record was performed on four consecutive days including one weekend day and at least one training day.

Before and after INT, the subjects carried out a performance test battery consisting of a standing long jump, an agility t-test and the Yo-Yo intermittent endurance test level 1 (Yo-Yo IE1) on a grass field. Prior to testing, the subjects refrained from severe physical activity for at least 48 h.

Within five days before and after the start of INT, the subjects arrived to the laboratory after an overnight fasting. Fasting blood samples were drawn from the antecubital vein and analysed for marker of health such as blood glucose and cholesterol. Body composition, including lean body mass (LBM), total fat mass (FM), regional fat mass, bone mineral content (BMC) and bone mineral density (BMD), was assessed by Dual-energy X-ray absorptiometry (DXA)

ELIGIBILITY:
Inclusion Criteria:

* age between 25-55 years
* less than two hours of physical training per week over the last two years before entering the study

Exclusion Criteria:

* biking for transportation more than 40 km/week
* diagnosed with severe diseases
* medical treatment with a documented effect on body composition
* abuse of alcohol/drugs
* pregnancy or breastfeeding.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2016-05-21 (Actual); Primary Completion 2016-11-25 (Actual); Study Completion 2016-11-25 (Actual)

PRIMARY OUTCOMES:
Lean body mass | 10 weeks
  Kg

SECONDARY OUTCOMES:
Bone density | 10 weeks
  g/cm2
Body fat percentage | 10 weeks
  % body weight

CONTACTS AND LOCATIONS:
Overall Officials: Jens Bangsbo, Dr. Sci, Study Chair — Department of Nutrition, Exercise and Sports
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No